CLINICAL TRIAL: NCT02981004
Title: PAR I - Prothesis-to-Annulus Relation (PAR) as Predictor of Hemodynamic Outcome in Aortic Valve Replacement
Brief Title: PAR I - Patient-to-Annulus Relation I
Acronym: PARI
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-09-015-GE-TV
Record Dates: First submitted 2016-10-21; First posted 2016-12-02 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Aortic Valve Disease
Keywords: Aortic valve disease, patient prosthesis mismatch
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Prosthesis-to-Annulus Relation I (PAR I) trial is a German multicenter study assessing the relation between the prosthetic GOA and the area of LVOT as potentially new parameter for the prediction of hemodynamic outcome. The results may possibly guide future valve size selection an may allow prediction of functionally relevant PPM (Patient-Prosthesis-Mismatch)

DETAILED DESCRIPTION:
Great debates revolve around the hemodynamic performance of prosthetic tissue valves. It is influenced by the design and the specific sizing strategy. Design determines the actual geometric orifice area (GOA), sizing strategy the actual size of the selected valve. Currently, hemodynamic performance is generally assessed by determining the effective orifice area (EOA, derived from the continuity equation by relating flow velocities and LVOT area). The question whether a prosthesis patient mismatch (PPM) is present is then addressed by relating EOA to body surface area (EOAi). However, this relation may not be reasonable because EOAi relates flow velocity twice to patient-specific anatomic parameters (LVOT area and body surface area) . Considering this potential methodological flaw, debate and confusion regarding PPM is easily understood, despite the fact that, intuitively leaving a gradient behind after aortic valve replacement cannot be irrelevant. Thus a reliable and comparable method to determine the presence of PPM is needed. In PAR I Trial the relation between true prothetic GOA and LVOT area will be assesses as a potentially new parameter for prediction of hemodynamic outcome, to possibly guide future valve size selection (inclusive valve-in-valve) and to allow the detection of functionally relevant PPM. In the trial it will be assessed how anatomic dimensions of patients and implanted valves relate to each other and whether they allow the prediction of hemodynamic outcome.

ELIGIBILITY:
Inclusion Criteria:1.Patient has an indication for primary, isolated aortic valve implantation 2. Patient is above 18 Years old 3. Patient has signed patient informed consent 4. foreseen implantation of an Epic, Epic supra or Trifecta valve 5. Patient has sinus rhythm

Exclusion Criteria:

1. Patient is younger than 18 years
2. Patient has active endocarditis
3. Patient is not able or does not want to participate on follow-up
4. Patient is pregnant or nursing
5. Surgical widening of outflow tract is planned
6. Left ventricular ejection fraction is smaller than 50%
7. Patient has a mitral valve or tricuspid valve insufficiency or stenosis bigger or equal Grade II

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with aortic valve disease selected for tissue valve implantation (routine care)
Sampling Method: Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
recording of hemodynamic outcome of a aortic valve in mutual dependence of anatomical facts on the basis of echocardiographic parameter | postprocedure before discharge (less than 30 days after implant)
  Echocardiographic evaluation of the anatomical facts e.g. Left ventricular outflow area

SECONDARY OUTCOMES:
Mortality 30 days after implant | 30 days
  Mortality
Morbidity 30 days after implant | 30 days
  Morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Doenst, M.D.Ph.D., Principal Investigator — Head of Cardiac surgery department
Locations (7):
- Germany (7):
  - Herzzentrum Dresden, Dresden
  - Asklepios St. Georg, Hamburg
  - Department of Cardiothoracic Surgery, Jena
  - Hospital Bogenhausen, Munich
  - Herz- und Kreislaufzentrum Rotenburg / Fulda, Rotenburg (Wümme)
  - Krankenhaus der Barmherzigen Brüder, Trier
  - University Hospital of Ulm, Ulm